CLINICAL TRIAL: NCT05225922
Title: Effect of Communication Partner Training Program for the Management of Persons With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LHR/21/1110 Fazaila Ehsan
Record Dates: First submitted 2021-12-29; First posted 2022-02-07 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Aphasia
Keywords: Aphasia; Post Stroke; Communication Partner Training
MeSH Terms: conditions — Aphasia | interventions — Language Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Communication Partner Training:The group will receive usual care in addition to a CPT program, which will consist of face-to-face education and counselling sessions, a manual and telephone support.
  Interventions: Behavioral: Communication Partner Training
- Comparison Group (Active Comparator): This group will receive usual speech therapy sessions.
  Interventions: Other: Usual Speech and language Therapy

INTERVENTIONS:
Behavioral: Communication Partner Training — This intervention aims to improve the language, communication, participation and overall quality of life of the Person with Aphasia.
  Arms: Experimental
Other: Usual Speech and language Therapy — This group will receive usual speech and language therapy session.
  Arms: Comparison Group

SUMMARY:
Communication Partner Training (CPT) is an evidence-based intervention that teaches communication partners (e.g., family members, friends, healthcare workers) how to best support conversation and interaction for a person with aphasia. It does not matter how mild or severe a person's aphasia is, they can be a good candidate for CPT as long as their communication partner is motivated and willing to adapt their communication style. The objective of this study is to see the effects of communication partner training for the management of persons with aphasia. A randomized controlled trial will be conducted. In total, 6 dyads will be randomly assigned to the intervention (CPT program) or usual care (control) group. Statistical Package for Social Sciences (SPSS) V 25. will be used for Data analysis. Results will be extracted. Conclusion will be made after comparing the pre and post treatment results on person with aphasia.

DETAILED DESCRIPTION:
Communication Partner Training (CPT) is an evidence-based intervention that teaches communication partners (e.g., family members, friends, healthcare workers) how to best support conversation and interaction for a person with aphasia. It does not matter how mild or severe a person's aphasia is, they can be a good candidate for CPT as long as their communication partner is motivated and willing to adapt their communication style. The objective of this study is to see the effects of communication partner training for the management of persons with aphasia. A randomized controlled trial will be conducted. In total, 6 dyads will be randomly assigned to the intervention (CPT program) or usual care (control) group. The intervention group received usual care in addition to a CPT program, which consisted of face-to-face education and counselling sessions, a manual and telephone support. Data will be collected at baseline, three months, and six months. The main outcome for caregivers will be using appropriate conversational skills that will be measured by the Conversational Skills Rating Scale (CSRS). Secondary outcomes for patients will be health-related quality of life that will be measured by the Quality of Life (QOL) Scale. To see the effective communication between patient and communication partner, Communicative Effectiveness Index (CETI) will be used.

ELIGIBILITY:
Inclusion Criteria:

* The participant's aphasia must be caused by stroke and to have occurred at least 12 months before the study takes place.
* The participant's aphasia could be of all degrees of severity (clinically assessed as mild, moderate, or severe on GCS).
* The participants with aphasia are required to be 18 years or older, living at home or planned to live at home after rehabilitation, and have no other speech or language impairments (such as severe dysarthria)
* Others have to communicate with the person with aphasia on a regular basis (at least once a week).

Exclusion Criteria:

The participants will be excluded if the persons with aphasia:

* Are diagnosed with dementia or any other known significant cognitive impairment.
* Have significant hearing or vision problems.
* Have known alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Conversational Skills | 6 Months
  Enhanced Communication skills in terms of attentiveness, expressiveness, coordination and composure. Skills ranging from Inadequate (1) to Excellent (5).
Quality of communication life | 6 Months
  Increased quality of communication life on quality of communication life scale , higher rating showing more positivity.

CONTACTS AND LOCATIONS:
Overall Officials: Fazaila Ehsan, PhD*, Principal Investigator — Riphah International University; Nazia Mumtaz, PhD, Study Director — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simmons-Mackie N, Raymer A, Armstrong E, Holland A, Cherney LR. Communication partner training in aphasia: a systematic review. Arch Phys Med Rehabil. 2010 Dec;91(12):1814-37. doi: 10.1016/j.apmr.2010.08.026. PMID 21112422
- [Background] Lock S, Wilkinson R, Bryan K, Maxim J, Edmundson A, Bruce C, Moir D. Supporting Partners of People with Aphasia in Relationships and Cconversation (SPPARC). Int J Lang Commun Disord. 2001;36 Suppl:25-30. doi: 10.3109/13682820109177853. PMID 11340791
- [Background] Kagan A, Black SE, Duchan FJ, Simmons-Mackie N, Square P. Training volunteers as conversation partners using "Supported Conversation for Adults with Aphasia" (SCA): a controlled trial. J Speech Lang Hear Res. 2001 Jun;44(3):624-38. doi: 10.1044/1092-4388(2001/051). PMID 11407567
- [Background] Chang HF, Power E, O'Halloran R, Foster A. Stroke communication partner training: a national survey of 122 clinicians on current practice patterns and perceived implementation barriers and facilitators. Int J Lang Commun Disord. 2018 Nov;53(6):1094-1109. doi: 10.1111/1460-6984.12421. Epub 2018 Aug 27. PMID 30151877
- [Background] Croteau C, McMahon-Morin P, Le Dorze G, Baril G. Impact of aphasia on communication in couples. Int J Lang Commun Disord. 2020 Jul;55(4):547-557. doi: 10.1111/1460-6984.12537. Epub 2020 May 13. PMID 32400928
- [Background] Johansson MB, Carlsson M, Sonnander K. Communication difficulties and the use of communication strategies: from the perspective of individuals with aphasia. Int J Lang Commun Disord. 2012 Mar-Apr;47(2):144-55. doi: 10.1111/j.1460-6984.2011.00089.x. Epub 2011 Oct 25. PMID 22369055